CLINICAL TRIAL: NCT00279747
Title: A One Year Double-blind Trial to Investigate the Efficacy and Safety of Meloxicam Oral Suspension 0.25mg/kg and 0.125 mg/kg Administered Once Daily in Comparison to Naproxen Oral Suspension 5mg/kg Administered Twice Daily in Children With Juvenile Rheumatoid Arthritis.
Brief Title: A One Year Double-blind Trial to Investigate the Efficacy and Safety of Meloxicam Oral Suspension in Juvenile Rheumatoid Arthritis (JRA/JIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107.208
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Arthritis, Juvenile Rheumatoid
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Meloxicam; Naproxen

INTERVENTIONS:
Drug: meloxicam 0.25 mg/kg
Drug: meloxicam 0.125 mg/kg
Drug: naproxen 10 mg/kg

SUMMARY:
A one year double-blind trial to investigate the efficacy and safety of meloxicam oral suspension 0.25 mg/kg and 0.125 mg/kg administered once daily in comparison to naproxen oral suspension 5 mg/kg administered twice daily in children with Juvenile Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Objective: In an international, multicenter, double-blind, randomized clinical trial we evaluated the short-term (3 months) and long term (12 months) efficacy and safety of two doses of meloxicam oral suspension compared with naproxen in children with oligo and polyarticular course juvenile idiopathic arthritis (JIA).

Methods: Children with active oligo or polyarticular course JIA, requiring therapy with an NSAID were eligible for this trial. Patients were randomly allocated to therapy with meloxicam oral suspension 0.125 mg/kg body weight in single daily dose, meloxicam 0.25 mg/kg body weight in single daily dose, or naproxen 10 mg/kg body weight in two daily doses. The trial drugs were administered in a double-blind, double-dummy design for up to 12 months. Response rates were determined according to the American College of Rheumatology Pediatric 30% definition of improvement (ACR Ped 30). Safety parameters were assessed by evaluation of the adverse events in the 3 groups.

Study Hypothesis:

The null hypothesis of interest is that the magnitude of response with regard to the primary endpoint is equivalent between the treatment groups. The alternative is that there is any difference (two-sided) between any of the treatment groups.

Comparison(s):

Naproxen oral suspension 10 mg/kg body weight.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients and inpatients aged 2 to 16 years
* Diagnosis of idiopathic arthritis of childhood by ILAR criteria:

  * Age of onset less than 16 years
  * Arthritis in one or more joints defined as swelling, or - if no swelling is present - limitation in range of joint movement with joint pain or tenderness, which is not due to primary mechanical disorders
  * Duration of the disease > 6 weeks
  * Type of onset of disease during the first 6 months classified as polyarthritis (5 joints or more; rheumatoid factor positive or negative), oligoarthritis (4 joints or fewer) or systemic arthritis
* Oligoarthritic, extended oligoarthritic or polyarthritic current course of disease
* Active arthritis as defined above of at least 2 joints
* At least 2 other abnormal variables of any of the 5 remaining core set parameters. The physician and the parent ratings must be at least 10 mm on a 100 mm VAS scale and the CHAQ score more than 0.
* Patients requiring therapy with NSAIDs, i.e., the patient fits into one of the following categories:

  * New onset patient
  * Patient in remission, but experiencing a flare and now requiring an NSAID
  * Patient with insufficient therapeutic effect (ITE) or intolerability to another NSAID (other than Naproxen) and now must be changed
* Written informed permission given by the parent(s) or the subjects legally authorised representative in accordance with local legislation and ICH GCP
* Active assent given by the patient if the child is capable of understanding the given information (applies to children who have reached an intellectual age of 7 years or greater)

Exclusion Criteria:

* Patients with systemic course of JRA (intermittent fever with or without rash or other organ involvement) or with current systemic involvement
* All rheumatic diseases not covered by the inclusion criteria
* Any finding indicating that the patient has a clinically significant other disease than JRA at the time of enrollment
* Patients with abnormal, clinically relevant laboratory values not related to their JRA
* Pregnancy or breast feeding
* Women of childbearing potential not using adequate contraception precaution: attention should be drawn to reports that NSAIDs were reported to decrease the effectiveness of intrauterine devices (R95-0164)
* History of bleeding disorders, gastrointestinal bleeding or cerebrovascular bleeding
* Active peptic ulcer within the last 6 months
* Treatment with more than one SAARD/DMARD (slow-acting antirheumatic drug/disease-modifying antirheumatic drug) during the last 3 months prior to study entry
* Change in treatment with SAARDs/DMARDs during the last 3 months prior to study entry or intended change during the trial duration
* Change in treatment with corticosteroids during the last month prior to study entry or intended change during the trial duration with exception of local therapy for uveitis
* One of the following therapies during the last 3 months prior to study entry or their intended use during the trial treatment period

  * Systemic treatment (except for intra-articular injections) with corticosteroids at a dose higher than 10 mg/day or 0.2 mg/kg/day (prednisone equivalent), respectively (whichever is lower)
  * Treatment with hydroxychloroquine at a dose higher than 10 mg/kg/day
  * Treatment with cyclosporine at a dose higher than 5 mg/kg/day
  * Treatment with methotrexate at a dose higher than 15 mg/m2/week
  * Treatment with other cytotoxic agents, gold compounds, D-penicillamine, Enbrel (etanercept), biologic agents and experimentals
* Intra-articular injections of corticosteroids during the last month prior to study entry and intended injections during the first 4 weeks of the trial treatment period
* Concomitant administration of other NSAIDs (including topical forms for skin with exception of local therapy for uveitis) or analgesic agents except paracetamol or acetaminophen

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 226
Dates: Start 2000-09; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Response rates according to ACR Ped 30 | after 12 weeks of treatment

SECONDARY OUTCOMES:
Global assessment of overall disease activity by investigator | up to 12 months
Parent global assessment of overall well-being | up to 12 months
Assessment of functional disability by means of Childhood Health Assessment Questionnaire (CHAQ) | up to 12 months
Number of joints with active arthritis | up to 12 months
Number of joints with limited range of motion | up to 12 months
Erythrocyte Sedimentation Rate (ESR) | up to 12 months
Parent global assessment of arthritis | up to 12 months
Parent global assessment of pain | up to 12 months
Children's assessment of discomfort | up to 12 months
Change in functional classification (Steinbrocker classification) | up to 12 months
Final global assessment of efficacy by parent | week 12, 12 months
Final global assessment of efficacy by investigator | week 12, 12 months
Withdrawals due to inadequate efficacy | up to 12 months
Paracetamol / acetaminophen consumption | up to 12 months
Final global assessment of tolerability by parent | week 12, 12 months
Final global assessment of tolerability by investigator | week 12, 12 months
Incidence and intensity of adverse events (AEs) | 12 months
Incidence of laboratory adverse events | 12 months
Withdrawal due to adverse event | 12 months
Duration of hospital stay due to gastrointestinal serious adverse event (GI-SAE) | week 12, 12 months
Duration of hospital stay due to adverse events related to trial drug administration | week 12, 12 months
Additional visits to a physician due to gastrointestinal adverse event (GI-AE) | week 12, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (34):
- Austria (3):
  - Landes-Kinderklinik Linz, Linz
  - Univ.-Klinik für Kinder- und Jugendheilkunde Wien, Vienna
  - Gottfried Preyersches Kinderspital d. Stadt Wien, Vienna
- Belgium (3):
  - UZ Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
  - Boehringer Ingelheim Investigational Site, Merksem
- France (6):
  - Boehringer Ingelheim Investigational Site, Angers
  - Boehringer Ingelheim Investigational Site, Lille
  - Boehringer Ingelheim Investigational Site, Marseille
  - Boehringer Ingelheim Investigational Site, Paris
  - Boehringer Ingelheim Investigational Site, Strasbourg
  - Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (6):
  - Rheumaklinik Bad Bramstedt GmbH, Bad Bramstedt
  - Neurologie, Bremen
  - Universität Erlangen, Erlangen
  - Martin-Luther-Universität Halle, Halle
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Bayrische Julius-Maximilians-Universität, Würzburg
- Italy (9):
  - Ospedale Meyer, Florence
  - Istituto G. Gaslini, Genova
  - Istituto Ortopedico Gaetano Pini, Milan
  - II Università degli Studi di Napoli, Napoli
  - Università Federico II, Napoli
  - Clinica Pediatrica I, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale Pediatrico Bambin Gesù, Roma
  - IRCCS Burlo Garofalo, Trieste
- Russia (4):
  - Institute of Rheumatology of RAMN, Moscow
  - Medical Faculty of Russian People Friendship University, Moscow
  - Scientific Research Institute of Pediatric Hematology, Moscow
  - Medical Academy Setchenov, Moscow
- United Kingdom (3):
  - Dept. of Child Health, London
  - Booth Hall Childrens Hospital, Manchester
  - Paediatric Department, Wolverhampton